CLINICAL TRIAL: NCT03959319
Title: Comparison of Movement Pattern Training and Manual Therapy for Prearthritic Hip Disorders: a Pilot Randomized Clinical Trial
Brief Title: Comparison of Movement Pattern Training and Manual Therapy for Prearthritic Hip Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Foundation for Physical Therapy, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201901005
Record Dates: First submitted 2019-05-20; First posted 2019-05-22 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Hip-related Groin Pain; Femoroacetabular Impingement; Dysplasia Mild; Prearthritic Hip Disorder
Keywords: clinical trial; rehabilitation; joint mobilization; movement training
MeSH Terms: conditions — Femoracetabular Impingement | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: Participants will complete self-report questionnaires and participate in a clinical examination that will include movement pattern, range of motion and quantitative sensory assessment. Participants will be randomized into one of two treatment groups, movement pattern training (MoveTrain) or manual therapy (ManTher). Both groups will participate in 10 supervised sessions within a 12 week time frame. MoveTrain will include task-specific training to optimize biomechanics during daily tasks and patient-specific tasks including work and fitness. ManTher will include select manual techniques including joint and soft tissue mobilization. Both groups will receive a home exercise program. At 13 weeks after enrollment, participants will return for testing to assess post-treatment improvements in primary and secondary outcomes. We also obtain 6 and 12 month questionnaires to assess patient outcomes.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The principle investigator and research staff who will be completing outcome assessments and measurements will be blinded to treatment group. Given the nature of the treatment, it is not possible to blind the care provider or the participant from the treatment group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Movement Pattern Training (Experimental): Focus will be on task-specific training to improve lower extremity movement patterns during basic daily tasks, such as sit to stand and stairs, and reported patient-specific tasks. Patient education will include instruction in abnormal movement patterns and methods to optimize movement patterns during each task. Tasks will be prioritized based on patient-report of activity limitations during the baseline examination. For example, during the first visit, the treating physical therapist will begin with the daily and patient-specific tasks that the patient reported as being most bothersome. Exercises will include repeated practice of functional tasks using optimized movement patterns. Based on the participant's performance, the difficulty of the task-specific activities will be progressed by varying the repetitions performed, increasing the load or changing the support surface. The home program will consist of repeated practice of tasks performed during the supervised sessions.
  Interventions: Other: Movement Pattern Training
- Manual Therapy (Joint Mobilization) (Active Comparator): Focus will be on reducing pain and improving pain-free range of motion using manual techniques provided by the physical therapist and exercise performed in the home program. Patient education will include instruction to the benefits of manual therapy and the proposed effects on pain and joint mobility. Joint mobilizations to be used with each patient will be prioritized based on the restrictions, defined as stiffness or pain that is limiting joint range of motion, noted on the patient's baseline examination. For example, during the first visit, the treating physical therapist will begin with the two most restricted motions noted in the baseline exam and perform a standard assessment to determine treatment parameters. The home program will include joint range of motion and stretching exercises to complement techniques performed during the supervised sessions.
  Interventions: Other: Manual Therapy

INTERVENTIONS:
Other: Movement Pattern Training — Treatment will include 10 supervised sessions over 12 weeks and instruction in a home exercise program After randomization, participants will be scheduled with a physical therapist trained in standard procedures. Treatment will include assessment of patient goals, patient education and instruction in a home program. Patient education will focus on patient-specific tasks, identified by the participant to be symptom-producing.
  Arms: Movement Pattern Training
Other: Manual Therapy — Treatment will include 10 supervised sessions over 12 weeks and instruction in a home exercise program After randomization, participants will be scheduled with a physical therapist trained in standard procedures. Treatment will include assessment of patient goals, patient education and instruction in a home program. Patient education will focus on patient-specific tasks, identified by the participant to be symptom-producing.
  Other Names: Joint Mobilization
  Arms: Manual Therapy (Joint Mobilization)

SUMMARY:
Significance: Intra-articular, prearthritic hip disorders (PAHD) result in substantial dysfunction in young adults and are proposed precursors to hip osteoarthritis (OA). Our long term goal is to develop effective treatment strategies for people with PAHD that will improve function, decrease pain and prevent or delay the onset of OA. The purpose of this study is to compare movement pattern training (MoveTrain) and manual therapy (ManTher) in their effect on post-treatment, patient-reported outcomes and targeted impairments thought to contribute to PAHD.

This pilot study will collect sufficient data to power a future study that will determine the efficacy of MoveTrain compared to ManTher for people with PAHD. Participants with PAHD will be randomized into one of two treatment groups, MoveTrain or ManTher. The Hip disability and Osteoarthritis Outcome Score (HOOS) will be the primary outcome measure. A measure of hip adduction motion during functional tasks and quantitative sensory assessment (pain pressure threshold and temporal summation) will be the secondary measures used to assess the effect of respective treatment on the impairments thought to contribute to PAHD, thus addressing the mechanisms of pain. Upon completion of this study, we will be positioned to implement a large RCT (randomized clinical trial) to definitively assess the efficacy of MoveTrain and ManTher to improve PAHD.

Specific Aims: To obtain preliminary estimates of effect sizes for planning the future definitive randomized clinical trial,

Aim 1 (Function): we will compare post-treatment improvements in hip-specific, patient-reported outcomes among the two treatment groups. After treatment completion:

Aim 2 (Mechanism): we will compare pre- and post-treatment measures in lower extremity movement patterns during functional tasks (MoveTrain) and quantitative sensory testing (ManTher). After treatment completion:

Aim 3 (Prognosis): we will determine the association among personal factors at baseline (demographic and psychosocial) and treatment prognosis (improvement in HOOS).

Impact: Our line of research will improve our understanding of each proposed treatment and its effect on patient function and each treatment's targeted impairment. This improved understanding will lead to the development of treatment strategies that will ultimately result in comparative effectiveness studies of surgical and non-surgical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years

  * Must be scheduled before their 40th birthday
* Have frequent hip joint symptoms, defined as pain, aching or stiffness within the hip joint for at least 3 months during the past 12 months
* Hip joint pain confirmed upon physical exam
* Report pain >= 3/10
* Reports functional limitation as demonstrated by modified Harris Hip Score <90
* Has protective sensation in the feet

Exclusion Criteria:

* Previous hip surgery, fracture, pelvic/hip infection or cancer
* Pain due to high impact trauma
* Inflammatory disease, e.g. rheumatoid arthritis, gout
* Acute pain in another joint that limits functional activities
* Perthes disease or slipped capital femoral epiphysis
* Hip pain referred from another source, e.g. lumbar spine
* Neurological involvement affecting balance or coordination
* Use of assistive gait device for more than 50% of time walking
* Pain, numbness or tingling in the lower extremity
* Pregnancy or given birth in previous 12 weeks
* Unwilling to refrain from taking NSAIDs 1-2 days prior to testing session
* Unable to attend regular physical therapy sessions
* Unable to complete 12 month follow up session

  * Avascular Necrosis
  * Ehler's Danlos Syndrome

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Function Using the Hip disability and Osteoarthritis Outcome Score Activities of Daily Living Subscale | Immediately after treatment (13 weeks after baseline)
  The Hip disability and Osteoarthritis Outcome Score (HOOS) is a hip-specific patient-reported outcome measure that has 5 subscales. Each subscale is score separately and ranges from 0-100, 100 = no disability, therefore higher values indicate a better outcome.
Change in Function Using the Hip disability and Osteoarthritis Outcome Score Symptom Subscale | Immediately after treatment (13 weeks after baseline)
  The Hip disability and Osteoarthritis Outcome Score (HOOS) is a hip-specific patient-reported outcome measure that has 5 subscales. Each subscale is score separately and ranges from 0-100, 100 = no disability, therefore higher values indicate a better outcome.
Percentage of Participants Who Are Adherent to Treatment Attendance | Immediately after treatment (13 weeks after baseline)
  Percentage of study participants who attend 90% (9/10) of the supervised treatment sessions.
Retention Rate | Immediately after treatment (13 weeks after baseline)
  Percentage of those enrolled at baseline who completed testing after treatment

SECONDARY OUTCOMES:
Home Exercise Program (HEP) adherence | Immediately after treatment (13 weeks after baseline)
  Participants were instructed to perform their HEP 5 times per week1 time per day. The variable for HEP adherence was calculated as the total number of days reported by the participant to have completed the prescribed exercises, summed over the entire treatment period, and divided by the total number of treatment days.
Patient treatment receipt | Immediately after treatment (13 weeks after baseline)
  The total number of exercises the physical therapist reviewed and the total number of those exercises they rated as independent were each summed across all treatment visits to derive the percent of exercises rated as independent across the entire treatment (Σ independent / Σ reviewed * 100).
Active ingredients for treatment delivery | Immediately after treatment (13 weeks after baseline)
  Treatment delivery assessed using chart reviews to determine if the active ingredients of the treatment was provided. The variable for treatment delivery is the proportion of active ingredients completed and documented by the treatment physical therapists for XX treatment visits
Change in hip adduction angle | Immediately after treatment (13 weeks after baseline)
  Change in hip adduction angle during functional tasks. Variable to assess movement pattern changes.
Change in hip adduction angle | On year after treatment completion
  Change in hip adduction angle during functional tasks. Variable to assess movement pattern changes.
Change in pain pressure threshold | Immediately after treatment (13 weeks after baseline)
  Pain pressure threshold is assessed with an algometer. This is a quantitative sensory testing to assess the patient's sensitivity to stimuli.
Change in pain pressure threshold | One year after treatment completion
  Pain pressure threshold is assessed with an algometer. This is a quantitative sensory testing to assess the patient's sensitivity to stimuli.
Change in Function Using the Hip disability and Osteoarthritis Outcome Score Pain Subscale | Immediately after treatment (13 weeks after baseline)
  The Hip disability and Osteoarthritis Outcome Score (HOOS) is a hip-specific patient-reported outcome measure that has 5 subscales. Each subscale is score separately and ranges from 0-100, 100 = no disability, therefore higher values indicate a better outcome.
Change in Function Using the Hip disability and Osteoarthritis Outcome Score Pain Subscale | One year after treatment completion
  The Hip disability and Osteoarthritis Outcome Score (HOOS) is a hip-specific patient-reported outcome measure that has 5 subscales. Each subscale is score separately and ranges from 0-100, 100 = no disability, therefore higher values indicate a better outcome.
Change in Function Using the Hip disability and Osteoarthritis Outcome Score Sport and Recreation Subscale | Immediately after treatment (13 weeks after baseline)
  The Hip disability and Osteoarthritis Outcome Score (HOOS) is a hip-specific patient-reported outcome measure that has 5 subscales. Each subscale is score separately and ranges from 0-100, 100 = no disability, therefore higher values indicate a better outcome.
Change in Function Using the Hip disability and Osteoarthritis Outcome Score Sport and Recreation Subscale | One year after treatment completion
  The Hip disability and Osteoarthritis Outcome Score (HOOS) is a hip-specific patient-reported outcome measure that has 5 subscales. Each subscale is score separately and ranges from 0-100, 100 = no disability, therefore higher values indicate a better outcome.
Change in Function Using the Hip disability and Osteoarthritis Outcome Score Quality of Life Subscale | Immediately after treatment (13 weeks after baseline)
  The Hip disability and Osteoarthritis Outcome Score (HOOS) is a hip-specific patient-reported outcome measure that has 5 subscales. Each subscale is score separately and ranges from 0-100, 100 = no disability, therefore higher values indicate a better outcome.
Change in Function Using the Hip disability and Osteoarthritis Outcome Score Quality of Life Subscale | One year after treatment completion
  The Hip disability and Osteoarthritis Outcome Score (HOOS) is a hip-specific patient-reported outcome measure that has 5 subscales. Each subscale is score separately and ranges from 0-100, 100 = no disability, therefore higher values indicate a better outcome.
Change in Function Using the Hip disability and Osteoarthritis Outcome Score Activities of Daily Living Subscale | One year after treatment completion
  The Hip disability and Osteoarthritis Outcome Score (HOOS) is a hip-specific patient-reported outcome measure that has 5 subscales. Each subscale is score separately and ranges from 0-100, 100 = no disability, therefore higher values indicate a better outcome.
Change in Function Using the Hip disability and Osteoarthritis Outcome Score Symptom Subscale | One year after treatment completion
  The Hip disability and Osteoarthritis Outcome Score (HOOS) is a hip-specific patient-reported outcome measure that has 5 subscales. Each subscale is score separately and ranges from 0-100, 100 = no disability, therefore higher values indicate a better outcome.
Change in movement evoked pain | Immediately after treatment (13 weeks after baseline)
  Movement evoked pain was assessed as a Numeric Pain Rating Scale (NPRS) after performance of a repetitive step down task and a repetitive deep squat task.
Change in movement evoked pain | One year after treatment completion
  Movement evoked pain was assessed as a Numeric Pain Rating Scale (NPRS) after performance of a repetitive step down task and a repetitive deep squat task.
Change in Function Using the International Hip Outcome Tool (iHOT-33) | Immediately after treatment (13 weeks after baseline)
  The iHOT is a hip-specific patient-reported outcome measure that represents the patient's report of symptoms, activity limitations, as well as emotional and social status. the score ranges from 0-100, 100 = no disability, therefore higher values indicate a better outcome.
Change in Function Using the International Hip Outcome Tool (iHOT-33) | One year after treatment completion
  The iHOT is a hip-specific patient-reported outcome measure that represents the patient's report of symptoms, activity limitations, as well as emotional and social status. the score ranges from 0-100, 100 = no disability, therefore higher values indicate a better outcome.
Change in Function Using the Patient Specific Functional Scale From Baseline to Post-treatment (13 Weeks) | Immediately after treatment (13 weeks after baseline)
  The Patient Specific Functional Scale (PSFS), a patient-reported outcome measure of patient-specific activity limitations. Patients are asked to identify "3-5 activities you are unable to do or having difficulties performing due to the pain or symptoms in your hip". Patients then rated level of difficulty from 0-10, 0 indicating they are unable to perform the activity and 10 indicating they are able to perform the activity at their preinjury level. The final score is an average of all scores provided. Change was calculated by subtracting the baseline PSFS from the post-treatment PSFS.
Change in Function Using the Patient Specific Functional Scale From Baseline to Post-treatment | One year after treatment completion
  The Patient Specific Functional Scale (PSFS), a patient-reported outcome measure of patient-specific activity limitations. Patients are asked to identify "3-5 activities you are unable to do or having difficulties performing due to the pain or symptoms in your hip". Patients then rated level of difficulty from 0-10, 0 indicating they are unable to perform the activity and 10 indicating they are able to perform the activity at their preinjury level. The final score is an average of all scores provided. Change was calculated by subtracting the baseline PSFS from the post-treatment PSFS.
Change in Average Pain Intensity Quantified by a Numeric Pain Rating Scale (NPRS) From Baseline to Post-treatment | Immediately after treatment (13 weeks after baseline)
  The numeric pain rating scale (NPRS) is a patient-reported outcome measure of pain intensity quantified using a 0-10 scale, 0 indicating the patient perceives no pain and 10 indicating the patient perceives the pain to be "worst pain imaginable". For average NPRS, patients are asked to rate what their pain was over the last week. Change was calculated by subtracting the baseline average NPRS from the post-treatment average NPRS.
Change in Average Pain Intensity Quantified by a Numeric Pain Rating Scale (NPRS) From Baseline to Post-treatment | One year after treatment completion
  The numeric pain rating scale (NPRS) is a patient-reported outcome measure of pain intensity quantified using a 0-10 scale, 0 indicating the patient perceives no pain and 10 indicating the patient perceives the pain to be "worst pain imaginable". For average NPRS, patients are asked to rate what their pain was over the last week. Change was calculated by subtracting the baseline average NPRS from the post-treatment average NPRS.
Change in Worst Pain Intensity Quantified by a Numeric Pain Rating Scale (NPRS) From Baseline to Post-treatment | Immediately after treatment (13 weeks after baseline)
  The numeric pain rating scale (NPRS) is a patient-reported outcome measure of pain intensity quantified using a 0-10 scale, 0 indicating the patient perceives no pain and 10 indicating the patient perceives the pain to be "worst pain imaginable". For worst NPRS, patients are asked to rate what was their worst (highest) level of pain was over the last week. Change was calculated by subtracting the baseline worst NPRS from the post-treatment worst NPRS.
Change in Worst Pain Intensity Quantified by a Numeric Pain Rating Scale (NPRS) From Baseline to Post-treatment | One year after treatment completion
  The numeric pain rating scale (NPRS) is a patient-reported outcome measure of pain intensity quantified using a 0-10 scale, 0 indicating the patient perceives no pain and 10 indicating the patient perceives the pain to be "worst pain imaginable". For worst NPRS, patients are asked to rate what was their worst (highest) level of pain was over the last week. Change was calculated by subtracting the baseline worst NPRS from the post-treatment worst NPRS.

CONTACTS AND LOCATIONS:
Locations (1):
- Program in Physical Therapy, Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abbott JH, Robertson MC, Chapple C, Pinto D, Wright AA, Leon de la Barra S, Baxter GD, Theis JC, Campbell AJ; MOA Trial team. Manual therapy, exercise therapy, or both, in addition to usual care, for osteoarthritis of the hip or knee: a randomized controlled trial. 1: clinical effectiveness. Osteoarthritis Cartilage. 2013 Apr;21(4):525-34. doi: 10.1016/j.joca.2012.12.014. Epub 2013 Jan 8. PMID 23313532
- [Background] Borrelli B. The assessment, monitoring, and enhancement of treatment fidelity in public health clinical trials. J Public Health Dent. 2011 Winter;71 Suppl 1:S52-63. PMID 21656954
- [Background] Chimenti RL, Frey-Law LA, Sluka KA. A Mechanism-Based Approach to Physical Therapist Management of Pain. Phys Ther. 2018 May 1;98(5):302-314. doi: 10.1093/ptj/pzy030. PMID 29669091
- [Background] Harris-Hayes M, Czuppon S, Van Dillen LR, Steger-May K, Sahrmann S, Schootman M, Salsich GB, Clohisy JC, Mueller MJ. Movement-Pattern Training to Improve Function in People With Chronic Hip Joint Pain: A Feasibility Randomized Clinical Trial. J Orthop Sports Phys Ther. 2016 Jun;46(6):452-61. doi: 10.2519/jospt.2016.6279. Epub 2016 Apr 26. PMID 27117727
- [Background] Harris-Hayes M, Holtzman GW, Earley JA, Van Dillen LR. Development and preliminary reliability testing of an assessment of patient independence in performing a treatment program: standardized scenarios. J Rehabil Med. 2010 Mar;42(3):221-7. doi: 10.2340/16501977-0505. PMID 20411216
- [Background] Harris-Hayes M, Mueller MJ, Sahrmann SA, Bloom NJ, Steger-May K, Clohisy JC, Salsich GB. Persons with chronic hip joint pain exhibit reduced hip muscle strength. J Orthop Sports Phys Ther. 2014 Nov;44(11):890-8. doi: 10.2519/jospt.2014.5268. Epub 2014 Oct 9. PMID 25299750
- [Background] Harris-Hayes M, Steger-May K, Koh C, Royer NK, Graci V, Salsich GB. Classification of lower extremity movement patterns based on visual assessment: reliability and correlation with 2-dimensional video analysis. J Athl Train. 2014 May-Jun;49(3):304-10. doi: 10.4085/1062-6050-49.2.21. PMID 24955621
- [Background] Harris-Hayes M, Steger-May K, van Dillen LR, Schootman M, Salsich GB, Czuppon S, Clohisy JC, Commean PK, Hillen TJ, Sahrmann SA, Mueller MJ. Reduced Hip Adduction Is Associated With Improved Function After Movement-Pattern Training in Young People With Chronic Hip Joint Pain. J Orthop Sports Phys Ther. 2018 Apr;48(4):316-324. doi: 10.2519/jospt.2018.7810. Epub 2018 Mar 16. PMID 29548270
- [Background] Hwang CT, Van Dillen LR, Haroutounian S. Do Changes in Sensory Processing Precede Low Back Pain Development in Healthy Individuals? Clin J Pain. 2018 Jun;34(6):525-531. doi: 10.1097/AJP.0000000000000563. PMID 29016389
- [Background] Moss P, Sluka K, Wright A. The initial effects of knee joint mobilization on osteoarthritic hyperalgesia. Man Ther. 2007 May;12(2):109-18. doi: 10.1016/j.math.2006.02.009. Epub 2006 Jun 13. PMID 16777467
- [Background] French HP, Cusack T, Brennan A, Caffrey A, Conroy R, Cuddy V, FitzGerald OM, Fitzpatrick M, Gilsenan C, Kane D, O'Connell PG, White B, McCarthy GM. Exercise and manual physiotherapy arthritis research trial (EMPART) for osteoarthritis of the hip: a multicenter randomized controlled trial. Arch Phys Med Rehabil. 2013 Feb;94(2):302-14. doi: 10.1016/j.apmr.2012.09.030. Epub 2012 Oct 16. PMID 23084955
- [Derived] DeMargel RD, Steger-May K, Haroutounian S, Zorn P, Cheng A, Clohisy JC, Harris-Hayes M. Personal factors and baseline function in patients undergoing non-operative management for chronic hip-related groin pain: a cross-sectional study. BMJ Open Sport Exerc Med. 2023 Nov 3;9(4):e001685. doi: 10.1136/bmjsem-2023-001685. eCollection 2023. PMID 37937305